CLINICAL TRIAL: NCT04729881
Title: Effects of Transcutaneous Electrical Nerve Stimulation, Ultrasound and Exercise on Pain, Functionality, Kinesophobia and Walking Speed in Individuals With Chronic Neck Pain
Brief Title: Effects of Exercise and Electrotherapy in Individuals With Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Sevda Yıldız, Physical Therapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 199400
Record Dates: First submitted 2021-01-21; First posted 2021-01-29 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The individuals are randomly allocated into control, intervention and specific exercise groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Rehabiliation Group (Experimental): Participants 5 days a week for 4 weeks; TENS, US and neck specific exercise program will be applied.
  Conventional TENS will be applied to the participants with the CefarCompex rehab400 (New Chattanooga Compex Rehab, USA) muscle rehabilitation device. It will be applied with electrodes coated with a special adhesive material for each participant for 20 minutes at a frequency of 60-120 Hz. In the study; 4 channels and 8 electrodes will be used. Electrodes will be placed paravertebrally in the cervicothoracic space, covering the painful area. The dose of the current will be increased as the patients become accustomed to the current intensity.
  Continuous Ultrasound will be applied to the participants due to chronic neck pain. It will be applied at a frequency of 1MHz and a dose of 1.5 W / cm2 for 5 minutes.
  Interventions: Other: Conventional Rehabiliation Group
- Spesific Exercise Group (Active Comparator): Participants will be given a home exercise program consisting of exercises specifically applied to the neck. Participants will be asked to practice the exercises 5 days a week. The application status of the participants' home exercise program will be followed by the researcher over the phone. Participants who do not practice the home exercise program will be excluded from the study. The exercise program to be applied to the participants in the exercise group is listed below.Cervical stretching exercise, Craniocervical flexion exercise, Neck isometric exercises, Cervical retraction exercise, Scapular retraction exercise, Modified push-up plus exercise.
  Interventions: Other: Spesific Exercise Group
- Control Group (Other)
  Interventions: Other: Control group

INTERVENTIONS:
Other: Conventional Rehabiliation Group — Transcutaneous Electrical Nerve Stimulation, Ultrasound and Exercise
  Arms: Conventional Rehabiliation Group
Other: Spesific Exercise Group — Cervical stretching exercise, Craniocervical flexion exercise, Neck isometric exercises, Cervical retraction exercise, Scapular retraction exercise, Modified push-up plus exercise
  Arms: Spesific Exercise Group
Other: Control group — No intervention will be aplied
  Arms: Control Group

SUMMARY:
In the treatment of neck pain, physiotherapy modalities such as ultrasound, Transcutaneous Electrical Nerve Stimulation (TENS), hot packs and personalized exercise approaches are frequently used. In this planned study, the effects of TENS, ultrasound and a program of stretching, posture and strengthening exercises on pain intensity, functionality, fear of movement and single-task and double-task walking speed in individuals with chronic neck pain will be investigated.

Participants will be evaluated initially and after four weeks.66 participants, who will be included in the study with more than 4 points from the neck disability questionnaire, will be randomly divided into 3 groups with 22 people in each group, regardless of the pain severity.Aches; With Visual Analogue Scale (VAS), their functionality; Kinesiophobia with Neck Disability Index; Single-task dual-task walking speeds with the Tampa Kinesiophobia Scale (TSK); It will be evaluated by the 10 Meter Walk Test.

DETAILED DESCRIPTION:
Among the musculoskeletal complaints of the spine, chronic neck pain (CKP), which is the second most common after low back pain, is seen in the society at a rate of 22-31%, and as it becomes chronic, it leads to an increase in doctor visits. KBA, which often originates from the spine and its surrounding soft tissues, can also be reflected from extravertebral tissues. Common clinical problems that cause neck pain include pathologies such as discopathies of cervical origin, spondylosis, stenosis, myofascial pain syndrome, and mechanical trauma caused by factors such as overuse and improper posture.It is known that being physically inactive in musculoskeletal system pain causes the pain to become chronic. However, CBA may prefer to remain physically inactive due to pain avoidance behaviors in individuals. Kinesiophobia, known as movement aversion; It is defined as "excessive avoidance of movement due to pain, re-injury and sensitivity". In addition to pain and impairment in functionality, CBA can lead to movement avoidance behaviors, many neuromuscular system and biomechanical disorders in individuals.In the studies in the literature, there are no studies that determine the effectiveness of the treatment approaches applied in individuals with CBA on functional status and pain, as well as movement avoidance and double-duty walking, which are effective in daily life. In this context, the aim of the study is to reveal the effectiveness of neck-specific exercises consisting of TENS, US and stretching-posture-strengthening exercises on pain intensity, functionality, kinesophobia and double and single task walking speed in individuals with CBA.

ELIGIBILITY:
Inclusion Criteria:

* Scoring over 4 points in the neck disability questionnaire,
* Having neck pain for at least 3 months,
* Agreeing to participate in the study voluntarily,
* 66 individuals between the ages of 18-65 will be included in the study.

Exclusion Criteria:

* Undergoing surgery in the cervical region,
* Having a history of acute trauma in the cervical region,
* Cervical vertebrae infection,
* Having a history of malignancy,
* Have inflammatory arthritis,
* Fracture, dislocation, tumor, infection,
* Who are pregnant,
* Receiving physical therapy within the last 1 year,
* With neurological deficits,
* Having a cardiac pacemaker,
* Patients with severe degeneration on magnetic resonance imaging will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Change between baseline and 4 weeks
  The scale used to determine the severity of pain is 100mm long, and its two ends are named differently on the vertical or horizontal line. The patient will be asked to mark a point on this line corresponding to the intensity of pain he / she feels.The distance between the marked point and the lowest end of the line (0 = no pain) will be measured in millimeters and the numerical value found will be recorded.
Neck Disability Index | Change between baseline and 4 weeks
  The Neck Disability Index scale, developed by Dr. Howard Vernon in 1980, was validated and reliable in 2012 by Kesiktaş et al. The scale evaluating the effects of neck pain on individuals' daily life activities consists of 10 titles: pain intensity, personal care, lifting, reading, headache, concentration, working, driving, sleeping and recreation. Individuals included in the study will be asked to score between 0 (no disability) and 5 (complete disability) for each title. The total score ranges from 0 (no disability) to 50 (complete disability). There is no 0-4 limitation in scoring the scale; 5-14: mild disability; 15-24: moderate disability; 25-34: Severe Disability; 35 and above are considered as Totally Disability.
Tampa Kinesiophobia Scale | Change between baseline and 4 weeks
  Developed to measure the fear of motion / re-injury, this scale includes the injury / re-injury and fear-avoidance parameters in work-related activities. 4-point Likert scoring (1 = Strongly disagree, 4 = Strongly agree) is used on the scale consisting of 17 questions. The Turkish validity and reliability of the scale has been proven. The person gets a total score between 17-68. The high score the person gets on the scale indicates that her kinesiophobia is also high.
10 Meter Walk Test | Change between baseline and 4 weeks
  It will be used to evaluate participants' single-task and double-task walking speed (Wa
  . The only task is to assess walking speed. In the ten-meter walking test, the person will be asked to walk at his / her own normal pace without speaking anything in the previously measured ten-meter field. The time will be started when the person's foot is on the starting line and will be terminated when they cross the finish line. Measurements will be recorded with the stopwatch in meters / second. To assess dual-task walking speeds; individuals will be asked to walk 2 counts from 100 during spontaneous walking of 10 meters and the measurements will be recorded in meters / second with a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Ataş Balcı, Assist.Prof, Study Director — Bahceşehir Unıversıty
Locations (1):
- Medamerikan medical center, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No